CLINICAL TRIAL: NCT04745871
Title: Diagnostic Performance of Prostate Specific Membrane Antigen (PSMA) Positron Emission Tomography/Computed Tomography (PET/CT) Imaging for Pre-operative Lymph Node Assessment in Intermediate and High-risk Non-metastasic Prostate Cancer.
Brief Title: Diagnostic Performance of PSMA PET/CT for Pre-operative Lymph Node Assessment in Intermediate and High-risk Non-metastasic Prostate Cancer (PREOP-PSMA ).
Acronym: PREOP-PSMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC20.0203
Record Dates: First submitted 2020-11-30; First posted 2021-02-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: TEP-PSMA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All patients with prostate cancer undergo PSMA PET/CT as part of the trial in addition to standard methods (abdo-pelvic MRI and a bone scan).
  Interventions: Diagnostic Test: PSMA PET/CT

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT — The PSMA PET/CT will be performed on an outpatient in the nuclear medicine department of the Brest University Hospital (CHRU). For this exam, the administration of 2-4 MBq/kg of 68Ga-HBED-CC-PSMA or 1,8-2,2 MBq/kg of 68Ga-PSMA-11 will be performed to patient by a single intravenous injection.

SUMMARY:
In France, prostate cancer is the most common cancer in men over 50 years of age (nearly 50,000 new cases per year) and is the second most common cause of cancer death in men (approximately 9,000 deaths per year). Although mortality has been declining since the end of the 1990s (about 7%/year), about 30 to 35% of them will have a biological recurrence.

Accurate assessment of local, regional and distant spread of the disease is therefore needed to design optimal personalised care for each patient, either curative or palliative.

Currently, in France, recommended disease assessment includes bone scintigraphy and Abdomino-Pelvic Magnetic Resonance Imaging. However, conventional imaging has limited performance with regard to lymph node extension.

Node dissection is the best way to assess node status. Currently, no imaging exam allows this level of accuracy.

Recently, molecular imaging has emerged as a promising tool to improve the initial extensional assessment of prostate cancer. Prostate-specific membrane antigen (PSMA) is a transmembrane glycoprotein, specific to the prostate, which is over-expressed on the surface of prostate cancer cells.

Recent studies of PSMA PET/CT as part of the initial extension assessment of prostate cancer report superior diagnostic performance in terms of sensitivity and specificity compared to conventional tests, as well as an impact of PSMA PET/CT on patient management.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer;
* Intermediate-risk prostate cancer (PSA level of 10- 20 ng/mL and/or Clinical tumor stage ≥ T2b and/or ISUP 2 or 3, AND with risk of lymph node extension > 5% according to the Briganti nomogram) or high-risk prostate cancer (PSA ≥ 20 ng/mL and/or TR ≥ T2c and/or ISUP 4 or 5) according to d'Amico classification;
* Curative treatment by radical prostatectomy chosen by the multidisciplinary consultation meeting.

Exclusion Criteria:

* Refusal or inability to participate in the study ;
* Low-risk prostate cancer according to D'Amico's classification, or an intermediate-risk but with a risk of lymph node extension <5% according to Briganti's nomogram;
* Curative treatment other than surgical treatment chosen;
* Life expectancy < 12 months;
* Karnofsky score < 70 or ECOG score > 2.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of PSMA PET/CT | Month 12
  The main objective of the trial is to determine the diagnostic performance of Positron Emission Tomography of Prostate Specific Membrane Antigen Ligands (PET-PSMA) for the detection of lymph node metastases in intermediate- and high-risk prostate neoplasia, whose radical treatment by prostatectomy is selected by the multidisciplinary consultation meeting.

SECONDARY OUTCOMES:
Impact of PSMA-PET in the surgical strategy of lymph node dissection. | Month 12
  To assess the impact of PSMA PET/CT in the surgical strategy of lymph node dissection, assessing the number of patients in whom lymph node dissection will be extended to a resectable PSMA-PET/CT suspicious area at the prostatic level.
Comparison of prostate tumor index lesion location on PSMA PET/CT and MRI with prostate histopathology after prostatectomy. | Month 12
  To compare MRI and PSMA PET/CT with histopathology at the prostate level (Pathological focal uptake detected on the 3 examinations (PSMA PET/CT and MRI vs. pathology = gold standard) for each of the 6 following prostate locations: base, middle, apex (right and left)).
Diagnostic performance of PSMA PET/CT for distant metastasis | Month 12
  To determine the positive predictive value of PSMA PET/CT to detect distant metastases in patients whose radical treatment by prostatectomy is selected by the multidisciplinary consultation meeting.
68Ga-HBED-CC-PSMA and et du 68Ga- PSMA-11 tolerance | Month 12
  The 68Ga-HBED-CC-PSMA tolerance and the et du 68Ga- PSMA-11 tolerance will be evaluated recording serious adverse events and adverse events during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.